CLINICAL TRIAL: NCT07277556
Title: Identification of Predictive Parameters for Developing a TURP Outcome Calculator for Preoperative Patient Assessment
Brief Title: TURP Outcome Prediction Calculator Study
Acronym: TURP-SCORE
Status: Not yet recruiting | Type: Observational
Sponsor: General Hospital Sveti Duh (Other)
Responsible Party: Principal Investigator, Adelina Hrkac, MD, FEBU, Principal Investigator, General Hospital Sveti Duh
Other Study IDs: KBSD-2025-03-3557; KBSD-URO--2025 (Registry Identifier: KB Sveti Duh Urology Institutional Research Registry)
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: BPH; LUTS; TURP; Uroflowmetry; IPSS; Outcome Prediction
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to identify which preoperative clinical, ultrasound, and uroflowmetry parameters can help predict the success of transurethral resection of the prostate (TURP) in adult male patients with symptomatic benign prostatic hyperplasia (BPH). The main questions it aims to answer are:

Which preoperative parameters (IPSS, prostate volume, post-void residual urine, Qmax, comorbidities) are associated with successful postoperative outcomes?

Can these parameters be used to develop a non-invasive calculator to estimate the likelihood of TURP success?

Participants will undergo routine clinical evaluation that is part of standard care, including:

* completion of the IPSS questionnaire
* digital rectal examination
* ultrasound measurement of prostate volume and residual urine
* uroflowmetry (Qmax and voided volume)
* standard laboratory testing Eligible participants will then undergo TURP as clinically indicated and return for postoperative assessments of symptom improvement and urinary flow parameters.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a common condition in aging men and may lead to lower urinary tract symptoms (LUTS), subvesical obstruction, and related complications such as urinary retention, bladder stones, recurrent infections, and renal impairment. Transurethral resection of the prostate (TURP) remains the standard surgical treatment for symptomatic benign prostatic obstruction (BPO). However, a subset of patients, particularly those with an underlying hypocontractile detrusor, may not benefit from TURP and continue to experience significant voiding dysfunction after surgery. Since formal urodynamic pressure-flow studies are invasive, time-consuming, and resource-intensive, there is clinical value in identifying non-invasive predictors of surgical success.

This prospective observational study will evaluate preoperative clinical, ultrasound, and uroflowmetry parameters associated with successful postoperative outcomes after TURP. Adult male patients with symptomatic BPH and an indication for TURP will undergo standardized assessment including medical history, IPSS questionnaire, digital rectal examination, serum PSA, ultrasound-determined prostate volume and post-void residual urine, and uroflowmetry parameters such as Qmax and voided volume. Comorbidities relevant to bladder function, including diabetes mellitus and neurological conditions, will be recorded. TURP will be performed according to standard clinical practice, and resected tissue will undergo routine histopathological evaluation.

Postoperative follow-up will include IPSS reassessment, uroflowmetry, and ultrasound measurement of residual urine at one month and during subsequent routine evaluations. Surgical outcomes will be categorized as successful or unsuccessful based on subjective symptom improvement and objective urinary flow parameters. Using the collected data, the study will identify which preoperative variables correlate with favorable postoperative outcomes. These parameters will subsequently be used to inform the development of a predictive TURP outcome calculator.

The anticipated value of this study is to support individualized clinical decision-making in patients with BPH, particularly those in whom the distinction between obstruction and impaired detrusor contractility is unclear. By identifying patients who are less likely to benefit from TURP based on non-invasive parameters, the resulting calculator may help reduce unnecessary procedures, avoid postoperative morbidity, and potentially limit the need for invasive urodynamic testing.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years or older
* Clinical diagnosis of benign prostatic hyperplasia (BPH)
* Indication for TURP based on symptoms or complications
* Completed preoperative evaluation (IPSS, ultrasound, PSA, uroflowmetry)
* Able to provide informed consent

Exclusion Criteria:

* Suspected or confirmed prostate cancer
* No clinical evidence of BPH
* Prior urodynamic diagnosis of underactive/neurogenic bladder
* Prior prostate surgery
* Inability to participate in follow-up

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Adult male patients with symptomatic benign prostatic hyperplasia undergoing clinically indicated transurethral resection of the prostate (TURP) at a single tertiary urology center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-13 (Estimated)

PRIMARY OUTCOMES:
Change in IPSS Score After TURP | 1 Month, 3 Months
  Improvement in lower urinary tract symptoms measured by the International Prostate Symptom Score (IPSS - validated questionnaire ranging from 0 to 35 points, where higher scores indicate more severe symptoms) one month after TURP compared to baseline.
Change in Qmax After TURP | 1 Month, 3 Months
  Improvement in maximum urinary flow rate (Qmax) measured by uroflowmetry after TURP
Change in Post-Void Residual Urine (PVR) | 1 Month, 3 Months
  Reduction in ultrasound-measured residual urine after voiding following TURP
Change in Voided Volume on Uroflowmetry | 1 Month, 3 Months
  Improvement in total voided volume after TURP

SECONDARY OUTCOMES:
Composite Surgical Success Rate | 1 Month, 3 Months
  Proportion of patients achieving predefined surgical success, based on combined improvements in IPSS, Qmax, voided volume, and post-void residual urine
Complication Rate Following TURP | 30 Days
  Frequency of postoperative complications categorized using Clavien-Dindo classification of surgical complications ranging from Grade 1 to Grade V (Grade 1 representing minor deviations from the normal postoperative course and Grade V representing patient death)

CONTACTS AND LOCATIONS:
Overall Officials: Adelina Hrkac, MD, Principal Investigator — Klinička bolnica "Sveti Duh", Zavod za urologiju

IPD SHARING:
Plan to Share IPD: No